CLINICAL TRIAL: NCT05495178
Title: Hepatobiliary Manifestations Following Two-Stages Elective Laparoscopic Restorative Proctocolectomy for Patients With Ulcerative Colitis. A Prospective Observational Study.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: hepatobiliary manifestations
Record Dates: First submitted 2022-08-06; First posted 2022-08-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hepatobiliary Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic restorative proctocolectomy — laparoscopic restorative proctocolectomy

SUMMARY:
Several studies using different methodological approach have revealed incomplete, old and conflicting data on the course of hepatobiliary manifestations after surgery. authors conducted a prospective observational study to evaluate the role of LRP on the course of hepatobiliary manifestations for a better knowledge of these manifestations that is necessary to improve their management.also, to evaluate the role of surgery on prevention of liver damage from progression of the disease.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) prevalence is expected to reach 1% of the population in many regions over the next decade. despite the fact that the primary clinical manifestations of IBD are centred in the gastrointestinal tract, 25-40% of IBD patients develop at least one extraintestinal manifestation (EIM).

Hepatobiliary manifestations constitute one of the most common EIMs in IBD . Hepatobiliary manifestations are much more commonly associated with ulcerative colitis (UC) and include primary sclerosing cholangitis (PSC), autoimmune hepatitis (AIH), fatty liver, cholelithiasis, primary biliary cholangitis, portal vein thrombosis, and hepatic abscess.

Most UC patients can be managed medically, but a minority requires proctocolectomy. Two-stage laparoscopic proctocolectomy (LPC) with ileal pouch-anal anastomosis (IPAA) is a cure for colitis, but its effect on hepatobiliary diseases is controversial.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18-69 years,
* both sex diagnosed as ulcerative colitis with at least one hepatobiliary manifestation
* underwent laparoscopic restorative proctocolectomy with ileal pouch anal anastomosis
* with or without gallstones.

Exclusion Criteria:

* age<18 years or > 69 years,
* alcohol abuse,
* pregnancy,
* severe heart failure or type II diabetes mellitus (defined as established diagnosis, HbA1c > 6.4%, non-fasting glucose level > 180 mg/dL, or on antidiabetic medication),
* development of complications or death related to the operation of LRP ,
* liver toxicity of IBD-related medications.,
* chronic viral hepatitis,
* haemochromatosis,
* Wilson's disease,

Ages: 18 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A prospective observational study was planned in our university hospitals' Surgical, internal and hepatology units on 167 patients with hepatobiliary manifestations in patients underwent one stage elective LRP for ulcerative colitis from June 2013 to June 2018. Inclusion criteria were all patients between 18-69 years, both sex diagnosed as ulcerative colitis with at least one hepatobiliary manifestation underwent laparoscopic restorative proctocolectomy with ileal pouch anal anastomosis with or without gallstones.indication for surgery in patients with UC was indicated according to ECCO guidelines on therapeutics in ulcerative colitis
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
severity of hepatobiliary manifestations after colectomy | 4 years
  severity of hepatobiliary manifestations are measured by abdominal ultrasonography,liver biopsy ,CT and MRCP

IPD SHARING:
Plan to Share IPD: Undecided